CLINICAL TRIAL: NCT03018587
Title: Feasibility Study of the TruSculpt Radiofrequency Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-16-TS12
Record Dates: First submitted 2017-01-09; First posted 2017-01-12 (Estimated); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Tissue Tightening

STUDY DESIGN:
Oversight: FDA-regulated Device: Yes

ARMS (1):
- All subjects (Experimental): All subjects will receive 1 truSculpt radiofrequency treatment in desired area.
  Interventions: Device: TruSculpt

INTERVENTIONS:
Device: TruSculpt — All subjects will receive 1 truSculpt radiofrequency treatment

SUMMARY:
A single-center, prospective, open-label feasibility study of the truSculpt radiofrequency device.

DETAILED DESCRIPTION:
A single-center, prospective, open-label study to evaluate the safety and efficacy of the Cutera truSculpt radiofrequency device for optimal delivery of thermal energy to the skin.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 18 to 70 years of age (inclusive)
2. Fitzpatrick Skin Type I - VI
3. Has visible fat bulges,skin laxity, or cellulite in the treatment area
4. Non-smoking for at least 6 months and willing to refrain from smoking for the duration of the study.
5. Subject must agree to not undergo any other procedure(s) in the treatment area during the study period.
6. Subject must be able to read, understand and sign the Informed Consent Form.
7. Subject must adhere to the follow-up schedule and study instructions.
8. Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes.
9. Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study, and no plans to become pregnant.

Exclusion Criteria:

1. Participation in a clinical trial of another device or drug in the target area during the study period.
2. Has a pacemaker, internal defibrillator, implantable cardioverter-defibrillator, nerve stimulator implant, cochlear implant or any other electronically, magnetically or mechanically activated implant.
3. Has metal implant(s) within the body that is local to the treatment area, such as surgical clips, plates and screws, intrauterine device (IUD), artificial heart valves or artificial joints.
4. Significant concurrent illness, such as diabetes mellitus, cardiovascular disease, peripheral vascular disease or pertinent neurological disorders.
5. Diagnosed or documented immune system disorders.
6. History of any disease or condition that could impair wound healing.
7. History of diseases stimulated by heat, such as recurrent herpes zoster in the treatment area, unless treatment is conducted following a prophylactic regimen.
8. Infection, dermatitis, rash or other skin abnormality in the target area.
9. Currently undergoing systemic chemotherapy or radiation treatment for cancer, or history of treatment in the target area within 3 months of study participation.
10. Pregnant or currently breastfeeding.
11. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ronan, M.D., Principal Investigator — Principal Investigator
Locations (1):
- Cutera Research Center, Brisbane, California, United States

IPD SHARING:
Plan to Share IPD: No
None. No individual participant data will be shared with other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Subjects
Started | 23
Completed | 19
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 4
Visible fat bulges, skin laxity, or cellulite [Count of Participants; unit: Participants] | 23

OUTCOME MEASURES:

1. Primary Outcome: Investigator Assessment of Improvement
Description: Degree of improvement in the treatment area at 12 weeks post-treatment compared with Baseline photo as assessed by the Investigator using Global Aesthetic Improvement Scale(GAIS): 4 = Very Significant Improvement (>75%), 3 = Significant Improvement (51 - 75%), 2 = Moderate Improvement (26 - 50%), 1 = Mild Improvement (5 - 25%), or 0 = No Change (<5%)
Time Frame: 12 weeks post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Subjects
Number analyzed (Participants) | 18
score on a scale | 0.67 (0.47)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 23/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=23)
Erythema (Skin and subcutaneous tissue disorders) | 21
Edema (Skin and subcutaneous tissue disorders) | 11
Nodules (Skin and subcutaneous tissue disorders) | 14 — Palpable firm lumps within subcutaneous fat developing 2-3 days after radiofrequency treatment in some areas treated which self-resolve typically within 4 to 8 weeks without intervention
Post treatment pain/discomfort (Skin and subcutaneous tissue disorders) | 6
Purpura (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/87/NCT03018587/Prot_SAP_000.pdf